CLINICAL TRIAL: NCT01782469
Title: A Prospective, Multi-center Study in Rheumatoid Arthritis Patients on Adalimumab to Evaluate Its Effect on Synovitis Using Ultrasonography in an Egyptian Population
Brief Title: Rheumatoid Arthritis Patients on Adalimumab to Evaluate Its Effect on Synovitis Using Ultrasonography in an Egyptian Population
Status: Terminated | Type: Observational
Why Stopped: Study stopped due to low enrollment
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-708
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Synovitis; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Synovitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis (RA) participants: Male or female participants at least 18 years of age with diagnosis of RA

SUMMARY:
This Post-Marketing Observational Study (PMOS) was conducted to assess the effectiveness of adalimumab on reducing synovitis (inflammation of the synovial membrane, which lines movable synovial joints, such as shoulders, elbows, wrists, knees, and hips) in adult participants with Rheumatoid Arthritis (RA) in Egypt. B-mode ultrasonography data was collected from participants receiving adalimumab treatment who had not been treated with any other anti-tumor necrosis factor (anti-TNF) therapy in the past.

DETAILED DESCRIPTION:
This study was a prospective, observational, single arm, multicenter study. Participants were treated with adalimumab in accordance with usual clinical care practices and local marketing authorization requirements. A total of 5 visits were planned: Baseline (Visit 1), Visits 2, 3, 4 and 5 (Week 13). The time interval between the baseline visit and the second visit was approximately 2-3 weeks, with a window of one week. Additional study objectives were to investigate the rate of RA progression via changes in the B-mode ultrasonography assessment score over time as well as changes in the number of joints with erosion over time. The study was terminated due to low enrollment.

ELIGIBILITY:
Inclusion Criteria:

A patient will be enrolled in this study if he/she fulfills ALL of the following criteria:

* Male or Female patients ≥ 18 years of age with diagnosis of RA
* Patient is eligible to start adalimumab therapy according to the local product label and prescription guidelines
* Patient is naïve to all biologics e.g. anti-cluster of differentiation 4 (anti-CD4) and anti-TNF treatments at the start of the study
* Patient has no history of inflammatory arthritis other than rheumatoid arthritis
* Patient has no history of lymphoma or leukemia or other malignancies
* Has negative result of tuberculosis (TB) screening test or is receiving TB prophylaxis as per local guidelines, Provided written Authorization to the investigator to use and/or disclose personal and/or health data, or Informed Consent if requested by the Local Regulations

Exclusion Criteria:

* Patients that are not diagnosed with rheumatoid arthritis as judged by the American College of Rheumatology criteria
* Patient is currently diagnosed with any condition other than rheumatoid arthritis that may affect radiography progression
* Susceptibility to infections including TB, as judged by the investigator
* Patient is carrier of Hepatitis B virus
* Patient is a pregnant or lactating female at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private clinics
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iman Ibrahim, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) Participants
Started | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Rheumatoid Arthritis (RA) Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Synovitis Measured by B-modal Ultrasonography Assessment Score After 13 Weeks of Treatment With Adalimumab.
Description: Synovitis was scored on a scale of 0 to 3 (0=none, 1=minor, 2=moderate, and 3=major presence). The sum of the scores of all 12 joints (elbow, wrist, second metacarpal (MCP), third MCP, knee and ankle) on both left and right sides is the ultrasonography assessment score, with a score range of 0-36.
Time Frame: Baseline (Visit 1) to 13 weeks
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis (RA) Participants
Number analyzed (Participants) | 15
units on a scale | -9.6 (4.98)

2. Secondary Outcome: Mean Percent Reduction in Ultrasonography Assessment Score
Description: Synovitis was scored on a scale of 0 to 3 (0=none, 1=minor, 2=moderate, and 3=major presence). The sum of the scores of all 12 joints (elbow, wrist, second metacarpal (MCP), third MCP, knee and ankle on both left and right sides) is the ultrasonography assessment score, with a score range of 0-36.
Time Frame: Baseline (Visit 1) to 13 weeks
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Rheumatoid Arthritis (RA) Participants
Number analyzed (Participants) | 16
Percent reduction
  Visit 2, n=16 | -20.99 (18.4)
  Visit 3, n=16 | -35.60 (25.36)
  Visit 4, n=16 | -48.42 (19.88)
  Visit 5, n=15 | -56.91 (24.81)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = 0.001, Wilcoxon signed-rank test — Mean percent reduction in ultrasonography assessment score at Vist 2 as compared to Baseline (Visit 1)
Statistical Analysis 2: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = 0.001, Wilcoxon signed-rank test — Mean percent reduction in ultrasonography assessment score at Vist 3 as compared to Baseline (Visit 1)
Statistical Analysis 3: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — Mean percent reduction in ultrasonography assessment score at Vist 4 as compared to Baseline (Visit 1)
Statistical Analysis 4: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = 0.001, Wilcoxon signed-rank test — Mean percent reduction in ultrasonography assessment score at Vist 5 as compared to Baseline (Visit 1)

3. Secondary Outcome: Mean Number of Joints With Detected Erosions
Description: A total of 12 joints (elbow, wrist, second metacarpal (MCP), third MCP, knee and ankle on both left and right sides) were assessed by ultrasonography at each study visit and the number of joints with erosion (wearing away) was documented.
Time Frame: Baseline (Visit 1) to 13 weeks
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Rheumatoid Arthritis (RA) Participants
Number analyzed (Participants) | 16
joints
  Visit 1, n=16 | 9.38 (1.89)
  Visit 2, n=16 | 8.69 (2.5)
  Visit 3, n=16 | 7.69 (3.3)
  Visit 4, n=16 | 6.75 (3.24)
  Visit 5, n=15 | 6.07 (2.91)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = .130, Wilcoxon signed-rank test — Mean number of joints with erosions at Vist 2 as compared to Baseline (Visit 1)
Statistical Analysis 2: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = 0.031, Wilcoxon signed-rank test — Mean number of joints with erosions at Vist 3 as compared to Baseline (Visit 1)
Statistical Analysis 3: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = 0.006, Wilcoxon signed-rank test — Mean number of joints with erosions at Vist 4 as compared to Baseline (Visit 1)
Statistical Analysis 4: Comparison: Rheumatoid Arthritis (RA) Participants; Test type: Superiority or Other; p = 0.003, Wilcoxon signed-rank test — Mean number of joints with erosions at Vist 5 as compared to Baseline (Visit 1)

4. Secondary Outcome: Percentage of Participants Who Achieved ≥ 20% Improvement in Both Tender Joint Count (TJC) and Swollen Joint Count (SJC)
Description: The American College of Rheumatology TJC and SJC was administered at each study visit. Participants were evaluated for tenderness and pain in 66 different joints when in motion (TJC), and 68 different joints were evaluated for swelling (SJC).
Time Frame: Baseline (Visit 1) to 13 weeks
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis (RA) Participants
Number analyzed (Participants) | 16
percentage of participants | 93.75 [80.4 to 107.1]

5. Secondary Outcome: Mean Change in Health Assessment Questionnaire (HAQ) Score
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥0.22. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5. Negative mean changes from Baseline in the overall score indicate improvement. Due to an error, HAQ data was not collected at 13 weeks.
Time Frame: Baseline (Visit 1) to 13 weeks
Population: Due to an error, HAQ data was not collected at 13 weeks. Therefore, only baseline data are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis (RA) Participants
Number analyzed (Participants) | 16
units on a scale | 1.19 (0.65)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time of informed consent until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment, up to 18 weeks.
Arm/Group | Rheumatoid Arthritis (RA) Participants
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.